CLINICAL TRIAL: NCT05900726
Title: Pilot Study to Determine Clinical Efficacy of Extracorporeal Pelvic Floor Magnetic Neuromuscular Stimulation in Patients With Faecal Incontinence.
Brief Title: Pelvipower for Faecal Incontinence
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Functional Gut Clinic (Other)
Responsible Party: Principal Investigator, Dr Anthony Hobson, Clinical Director, The Functional Gut Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FGC-20-001
Record Dates: First submitted 2023-01-31; First posted 2023-06-13 (Actual); Last update posted 2023-06-13 (Actual); Status verified 2023-06

CONDITIONS: Faecal Incontinence
MeSH Terms: conditions — Encopresis

STUDY DESIGN:
Intervention Model Description: This protocol describes a single blinded, two-armed, parallel-group, randomised exploratory study with control arm, assessing the effect of pelvic floor magnetic neuromuscular stimulation (Pelvipower) versus sham stimulation, in patients with faecal incontinence.
Who Masked: Participant
Masking Description: Randomised allocation to treatment or sham arm will be performed using sealedenvelope.com, the software will only be available to the study team. Participant ID's will be entered 001 - 036 randomisation tool on sealedenvelope.com where they will be assigned to group A (treatment) or group B (sham). A randomisation log will be kept in the site file. Participants will be blinded to which group they have been assigned too.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pelvipower chair (Experimental)
  Interventions: Diagnostic Test: High Resolution Anorectal Manometry; Diagnostic Test: Endoanal Ultrasound; Other: Bowel diary; Other: MYMOP2; Other: FIQOL; Other: FISI; Other: Follow up call; Other: St Mark's incontinence score
- Sham stimulation (Sham Comparator)
  Interventions: Diagnostic Test: High Resolution Anorectal Manometry; Diagnostic Test: Endoanal Ultrasound; Other: Bowel diary; Other: MYMOP2; Other: FIQOL; Other: FISI; Other: Follow up call; Other: St Mark's incontinence score

INTERVENTIONS:
Diagnostic Test: High Resolution Anorectal Manometry — A test used to measure the strength of the muscles in the anal canal
Diagnostic Test: Endoanal Ultrasound — An examination of the anal canal (back passage) that allows us to see the muscles involved in passing stool and the tissues that surround these.
Other: Bowel diary — A daily diary to assess episodes of faecal incontinence
Other: MYMOP2 — Questionnaire to assess individual symptoms, general wellbeing and activity in faecal incontinence
Other: FIQOL — Questionnaire to assess the quality of life with faecal incontinence
Other: FISI — Questionnaire to assess the severity of faecal incontinence
Other: Follow up call — At 28 days and 3 months post final pelvipower or sham session to assess faecal incontience after study period
Other: St Mark's incontinence score — A score of incontinence

SUMMARY:
Faecal incontinence (FI) is a common condition which drastically reduces patient's quality of life and for which there are few effective treatments. The causes of FI are multiple and include disturbances in neuromuscular function (and structure) of the anal canal, rectum and pelvic floor. Treatment options include antidiarrheals, laxatives, biofeedback, surgery, SNS and PTNS. This study will test the Pelvipower extracorporeal magnetic stimulation device as a treatment for faecal incontinence.

DETAILED DESCRIPTION:
First line treatment with antidiarrheal or laxative therapy can fail, and then it is common practice to employ biofeedback and physiotherapy techniques as second line conservative management strategies with the aim of improving muscle strength, sensory awareness and effective toileting technique, which in turn helps to reduce FI episodes . Whilst these techniques can be effective, a significant proportion of patients remain symptomatic and are then considered for potential surgical treatment.

Surgical treatment of FI can involve improving the structural integrity of the anal sphincter with a repair procedure, or via implantation of an electrical neurostimulator (sacral nerve stimulation - SNS). SNS has been shown to be effective in treating FI, but the procedure is invasive and expensive.

Percutaneous tibial stimulation (PTNS) is an intermediate treatment which involves stimulating the nerves on the top of the foot which project to the same spinal regions as those influenced through SNS. This requires patients to attend an outpatient clinic for up to 12 sessions, each lasting around 30-45 minutes. Stimulation is delivered via needle electrodes which connect to a stimulation device. A course of treatment costs approximately £2000 per patient for 1-year of treatment.

Whilst SNS and PTNS utilise electric neural stimulation, an alternative approach is through the use of magnetic stimulation as a way of activating neural pathways and inducing neuromuscular recovery. The technique is thought to work on the nerves and muscular structures in the anal canal. This technique has been employed in a broad range of disorders. Magnetic stimulation has some advantages as it can be delivered completely non-invasively using different sized magnetic coils placed over the region of interest.

Pelvipower (PonteMed AG, Switzerland) extracorporeal magnetic stimulation device built into a patient friendly chair, incorporating a rapid rate magnetic stimulation system through a stimulation coil. The coil can be used to non-invasively stimulate the nerves and muscles in the pelvic floor that contribute to continence, and it has several potential advantages over existing techniques in terms of cost and convenience, with 6-12 weekly 15 minute sessions currently normal practice. Pelvipower has been used successfully in patients with urinary incontinence, but thus far little research exists in terms of its effect in treating faecal incontinence. However, one study of extracorporeal magnetic stimulation applied via a similar chair apparatus demonstrated increased muscle function in the anal canal, as well as a significant decrease in faecal incontinence. Although faecal incontinence was shown to improve in participants, the study did not include a sham treatment comparison group. The aim of this study is to evaluate the effect of the extracorporeal magnetic stimulation on faecal incontinence, using the Pelvipower© chair compared to a sham treatment.

ELIGIBILITY:
Inclusion Criteria:

1. >18 years of age
2. Female
3. Have suffered from faecal incontinence, for >6 months, sufficiently severe enough to warrant intervention . Previous exposure to treatment is not a contraindication to this.
4. Body Mass Index between 18.9 and 40.0kg/m2 (bounds included)
5. >6 months post-natal
6. ≥4 FI episodes during 2 week screening period

Exclusion Criteria:

1. Neurological disease which may affect continence (i.e. diabetic neuropathy, multiple sclerosis, Parkinson's disease etc)
2. Thromboses
3. Suffering from or recovering from a serious illness or operation
4. Faecal incontinence secondary to impaction
5. Currently using rectal irrigation
6. Currently undergoing biofeedback therapy
7. Pregnancy
8. Pacemaker in situ
9. Indwelling metal implants
10. Recent skeletomuscular injury or surgery in the last month
11. Congenital anorectal disorders such as cloacal defect
12. Participant has a > grade 2 rectal prolapse
13. Absence of native rectum due to surgery (anterior resection)
14. Previous anal/rectal surgery in the past 12 months
15. Stoma in situ
16. Chronic bowel diseases with chronic uncontrolled diarrhoea
17. Unable to discontinue Loperamide during washout period
18. Severe cardiac arrhythmia
19. Epilepsy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
Bowel diary - total FI episodes | up to 10 weeks
  Assessment of change in total faecal incontinence episodes as measured as a reduction by >= 50%

SECONDARY OUTCOMES:
Bowel diary - passive FI episodes | up to 10 weeks
  Assessment of change in passive faecal incontinence episodes as measured as a reduction by >= 50%
Bowel diary - urgency FI Episodes | up to 10 weeks
  Assessment of change in urge faecal incontinence episodes as measured as a reduction by >= 50%
St Mark's incontinence score | up to 5 months
  Effect of extracorporeal magnetic stimulation using the Pelvipower chair on FI, assessed using mean change from randomisation visit to post treatment visit FI scores (as measured by St Marks incontinence score) between treatment and sham groups.
Loperamide use | up to 10 weeks
  Mean change in loperamide use from randomisation to post- treatment visit between treatment and sham groups, measured using pre-treatment and post-treatment bowel diaries.
Measure Yourself Medical Outcome Profile 2 (MYMOP2) | up to 5 months
  Mean change from randomisation visit to post-treatment visit in questionnaire total score between treatment and sham groups.
Faecal incontinence quality of life questionnaire (FIQL) | up to 5 months
  Mean change from randomisation visit to post treatment visit in FIQOL score between treatment and sham groups.
Faecal incontinence symptom index (FISI) | up to 5 months
  Mean change from randomisation visit to post treatment visit in FISI score between treatment and sham groups.

OTHER OUTCOMES:
Assessment of anal canal resting tone | up to 10 weeks
  A) Mean change from randomisation visit to post treatment in mean anal resting pressure between treatment and sham groups. Measured using high resolution anorectal manometry, measured in mmHg.
Assessment of voluntary anal squeeze pressures | up to 10 weeks
  Mean change from randomisation visit to post treatment in mean voluntary squeeze pressure between treatment and sham groups - using high resolution anorectal manometry, measured in mmHg.
Assessment of rectal sensation | up to 10 weeks
  C) Mean change from randomisation visit to post treatment in rectal sensation thresholds (first constant sensation volume, urge to defecate volume and maximum tolerable volume) between treatment and sham groups, using balloon sensation testing as part of anorectal manometry. Thresholds measures of vol of air in balloon (ML) when sensations are noted by the participant.
Assessment of anal sensation | up to 10 weeks
  Mean change from randomisation visit to post treatment in anal sensitivity between treatment and sham groups. Measured using anorectal manometry and specialised anal sensitivity probes.

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Hobson, Principal Investigator — The Functional Gut Clinic
Locations (1):
- The Functional Gut Clinic, London, United Kingdom